CLINICAL TRIAL: NCT05255952
Title: EpiCANS : Epicardial Stimulation of the Cardiac Autonomic Nervous System
Brief Title: Epicardial Stimulation of the Cardiac Autonomic Nervous System
Acronym: EpiCANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC21_8946_04_EpiCANS
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Insufficiency
Keywords: cardiac plexus; Electrical stimulation
MeSH Terms: conditions — Heart Failure | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): 3 cycles of electrical stimualtions will be done at the end of cardiac surgery, before end of surgery (patient closure), under anaesthesia.
  Cardiac outcomes will be monitored
  Interventions: Procedure: Electrical stimulation

INTERVENTIONS:
Procedure: Electrical stimulation — Electrical stimulation of the cardiac plexus

SUMMARY:
The objective of the EpiCANS study is to evaluate the technique of stimulation of the cardiac autonomic nervous system (SNAC) directly at the epicardial level in humans during heart surgery.

Proof of concept study

DETAILED DESCRIPTION:
Isolated stimulation of the parasympathetic system induces a protective effect on long-term cardiac remodeling, but at the cost of inhibiting the sympathetic system. The role of the sympathetic system is to increase cardiac output in cases of acute heart failure.

Electrical stimulation of the cardiac plexus directly at the level of the heart allows simultaneous stimulation of the sympathetic and parasympathetic systems, whose complementary and not automatically antagonistic role is now recognized. Thus, direct stimulation of the plexus would optimize cardiac function in the short and long term by instantly improving cardiac output and decreasing pulmonary resistance as described in dogs by Kobayashi et al.

The objective of the EpiCANS study is to evaluate this technique in humans during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective cardiac surgery for valvular or coronary surgery
* Having received written and oral information about the protocol and having signed a written informed consent
* Affiliated or beneficiary of a social security plan

Exclusion Criteria:

* Patient with an indication for cardiac surgery:
* Urgent or semi-urgent
* Aortic surgery
* Heart transplantation
* Mechanical circulatory assistance
* Patients who have already undergone cardiac surgery
* Adults under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty, pregnant or breastfeeding women, minors, persons unable to express their consent, persons hospitalized for a different reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Variation of cardiac output | 15 min
  Cardiac output (milliliter per minute) before and after stimulation

SECONDARY OUTCOMES:
Variation of Cardiac rythm | 15 min
  Heart rate (beat per minute) before and after stimulation
Variation of aortic pressure | 15 min
  Aortic pressure (millimeter of mercury) before and after stimulation
Variation of pulmonary artery pressure | 15 min
  Pulmonary artery pressure (millimeter of mercury) before and after stimulation
Variation of central venous pressure | 15 min
  Central venous pressure (millimeter of mercury) before and after stimulation
Presence of atrial fibrillation | 15 min
  Atrial fibrillation related to stimulation
Adverses events | 10 days
  Advserse events during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Karl BOU NADER, Dr, Study Director — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No